CLINICAL TRIAL: NCT05755516
Title: Efficacy and Safety of the Self-expanding Intracranial Stent (Tonbridge) for Endovascular Treatment of Intracranial Aneurysms: A Prospective, Multi-center, Randomized, Open, Parallel Positive Controlled, Non-inferiority Trial
Brief Title: Efficacy and Safety of the Self-expanding Intracranial Stent (Tonbridge) for Endovascular Treatment of Intracranial Aneurysms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ton-Bridge Medical Tech. Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZHTQ202202
Record Dates: First submitted 2023-02-21; First posted 2023-03-06 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Self-expanding Intracranial Stent (Tonbridge)
  Interventions: Device: Self-expanding Intracranial Stent (Tonbridge)
- control group (Active Comparator): LVIS and LVIS Jr. (MicroVention)
  Interventions: Device: LVIS and LVIS Jr. (MicroVention)

INTERVENTIONS:
Device: Self-expanding Intracranial Stent (Tonbridge) — Stent assisted coiling with Self-expanding Intracranial Stent (Tonbridge).
  Arms: experimental group
Device: LVIS and LVIS Jr. (MicroVention) — Stent assisted coiling with LVIS and LVIS Jr. (MicroVention).
  Arms: control group

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Self-expanding Intracranial Stent (Tonbridge), by comparing the data obtained from Self-expanding Intracranial Stent (Zhuhai Tonbridge Medical Tech. Co., Ltd.) and LVIS/LVIS Jr. (MicroVention Europe SARL) for endovascular treatment of intracranial aneurysms.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, open, parallel positive controlled, non-inferiority trial. This clinical trial is conducted at more than 2 centers in China, and patients who intend to be treated with stent-assisted coiling for intracranial aneurysms are enrolled. Eligible patients are randomized into experimental group using Self-expanding Intracranial Stent (Tonbridge) or control group using LVIS and LVIS Jr. (MicroVention) in a 1:1 ratio. The purpose of this study is to evaluate the effectiveness and safety of the Self-expanding Intracranial Stent (Tonbridge).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years, any gender;
* Diagnosed as intracranial aneurysm and the subject is assessed as suitable for stent-assisted coiling;
* Subject or guardian is able to understand the purpose of study, shows sufficient compliance with the study protocol and provides a signed informed consent form.

Exclusion Criteria:

* Aneurysm rupture within 30 days before enrollment;
* Diagnosed as blood blister-like aneurysm, pseudoaneurysm, infected aneurysm, or aneurysm related to arteriovenous malformations;
* Conditions that are not appropriate for stent delivery and deployment judged by investigators (severe stenosis of parent artery, severe tortuosity of parent artery, stent failing to reach the lesion, stent in the target lesion of parent artery, etc.);
* Modified Rankin Scale (mRS) score ≥3;
* Heart, lung, liver and renal failure or other severe diseases (intracranial tumor, systemic infection, disseminated intravascular coagulation, myocardial infarction within 12 months before enrollment, history of severe psychosis, severe stenosis or occlusion of cerebral feeding artery, etc.);
* Major surgery within 30 days before enrollment；
* Known coagulation dysfunction or contraindication to anticoagulant and antiplatelet therapy;
* Known allergy to nickel-titanium alloy metal materials;
* Life expectancy <12 months;
* Pregnant or breastfeeding women;
* Subject has participated in other drug or medical device clinical trials within 1 month before signing informed consent;
* Other conditions judged by the investigators as unsuitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Successful occlusion rate of aneurysms at 6 months | 6 months±30 days post-procedure
  Successful occlusion is defined as complete occlusion or neck remnant (Raymond-Roy class I or Ⅱ), which is diagnosed by cerebrovascular DSA at 6 months post-procedure.

SECONDARY OUTCOMES:
Device success rate | intra-procedure
  Device success is that the stent is delivered to the target vessel successfully and covers the aneurysm neck effectively without stent migration or misplacement, etc. Device success is diagnosed by intraoperative cerebrovascular DSA.
Immediate successful occlusion rate of aneurysms | intra-procedure
  Successful occlusion is defined as complete occlusion or neck remnant (Raymond-Roy class I or Ⅱ), which is diagnosed by intraoperative cerebrovascular DSA.
Recurrence rate of aneurysms at 6 months | 6 months±30 days post-procedure
  Recurrence is defined as increased contrast agent filling into the aneurysm sac at post-operative review compared to immediate post-procedure.
Retreatment rate | 180±30 days, 360±30 days post-procedure
  Retreatment is defined as during the study period any additional treatment of the target aneurysm after the original procedure.
Operation satisfaction rate | intra-procedure
  The 5-point Likert scale is used to evaluate the operation satisfaction from three aspects: push performance, retracting performance and release performance. "Operation satisfaction rate" is defined as the proportion of investigational devices or comparators with Likert score≥12 points.
Incidence of parent artery stenosis (>50%) in target area | 180±30 days, 360±30 days post-procedure
  Parent artery stenosis in target area is defined as stenosis degree >50%, which is diagnosed by postoperative cerebrovascular DSA at 6 months, CTA or MRA at 12 months.
Incidence of parent artery occlusion in target area | 180±30 days, 360±30 days post-procedure
  Parent artery occlusion in target area is diagnosed by postoperative cerebrovascular DSA at 6 months, CTA or MRA at 12 months.
Incidence of stroke | 30±7 days, 360±30 days post-procedure
  Stroke includes hemorrhagic stroke and symptomatic ischemic stroke.
All-cause mortality | 30±7 days, 360±30 days post-procedure
  "All-cause mortality" is the proportion of subjects who die due to any cause.
Incidence of adverse events | 180±30 days, 360±30 days post-procedure
  "Incidence of adverse events" is the proportion of subjects with adverse events using the investigational device or the comparator.
Incidence of serious adverse events | 180±30 days, 360±30 days post-procedure
  "Incidence of serious adverse events" is the proportion of subjects with serious adverse events using the investigational device or the comparator.
Incidence of device deficiency | intra-procedure, 180±30 days post-procedure
  Device deficiency is the unreasonable risk that may endanger human health and life safety in the normal use of medical devices during clinical trials, such as labeling errors, quality problems and malfunctions.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, Principal Investigator — Changhai Hospital; Chuanzhi Duan, Principal Investigator — Southern Medical University, China
Locations (14):
- China (14):
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Zhuhai People's Hospital, Zhuhai, Guangdong
  - Tongji Hospital Tongji Medical College of HUST, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - General Hospital of Eastern Theater Command, Nanjing, Jiangsu
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Sichuan Academy of Medical Sciences·Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Changhai Hospital of Shanghai, Shanghai